CLINICAL TRIAL: NCT04507867
Title: Effect of a Nutritional Support System to Reduce Complications in Patients With Covid-19 and Comorbidities in Stage III
Brief Title: Effect of a NSS to Reduce Complications in Patients With Covid-19 and Comorbidities in Stage III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anahuac University (Other)
Responsible Party: Principal Investigator, Fernando Leal-Martinez, Doctor in Clinical Nutrition, Anahuac University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 202036
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: COVID19; Diabetes Mellitus; Hypertension; Obesity; Overweight; Oxygen Saturation; Mortality; Inflammation
Keywords: COVID19; Nutritional support; SARS-COV-2; Pneumonia; Supplementation; Probiotics
MeSH Terms: conditions — COVID-19; Diabetes Mellitus; Hypertension; Obesity; Overweight; Inflammation; Pneumonia

STUDY DESIGN:
Intervention Model Description: exploratory study, it is a controlled, blinded, randomized clinical trial design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: blinding was planned for patients and evaluators (treating physicians , care provider and laboratory personnel)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): Patients who received the standard diet
  Interventions: Other: Conventional nutritional support designed by hospital nutritionists
- Intervention group (Experimental): Patients who received the nutritional support system (NSS) and the standard diet
  Interventions: Dietary Supplement: Nutritional support system (NSS); Other: Conventional nutritional support designed by hospital nutritionists

INTERVENTIONS:
Dietary Supplement: Nutritional support system (NSS) — 1. Combination of three B vitamins (B1, B6 and B12) "Neurobion" 10 mg solution for IM injection, One every 24 hours for the first 5 days.
  2. Probiotics Saccharomyces boulardii CNCM I-745 "Floratil". One morning and one evening 250 mg capsule during the first 6 days
  3. One envelope of NSS-1 in the morning and one envelope in the afternoon mixed with 400 ml of water each, contain nutritional support system.
  Arms: Intervention group
Other: Conventional nutritional support designed by hospital nutritionists — Diet designed by the nutrition department according to comorbidities and intubation probability. Food will be established according to the provisions of the ISSEMYM Toluca Arturo Montiel Rojas Medical Center.

SUMMARY:
The disease caused by SARS-CoV-2, has derived a pandemic in which its evolution and complications depend on the immune capacity of the host. The virus has been characterized by presenting an inflammatory cascade, increased by the overproduction of proinflammatory cytokines, the decrease in metalloenzymes and also the rapid spread of the virus. There are several lines of treatment, however, nutritional treatment only considered a caloric intake. For this reason, this study will evaluate the evolution of patients with COVID-19 assisted by nutritional support system and the effect of this therapy in reducing complications and comorbidities.

Research question: Will the nutritional support system reduce complications in stage III positive COVID-19 patients with comorbidities (type 2 DM, SAH, overweight / obesity with BMI <35), with a better benefit than that achieved with the conventional nutritional treatment ?.

Hypothesis: The nutritional support system will reduce the complications of patients with COVID-19 in stage III with comorbidities. General Objective: To determine the effect of the use of a nutritional support system on complications in patients with COVID-19 in stage III with comorbidities.

Methodology: A controlled, blinded, randomized clinical trial will be conducted in patients with COVID-19, hospitalized at the ISSEMYM Toluca Arturo Montiel Rojas Medical Center, who meet the inclusion criteria. The evolution of the group of patients receiving the nutritional support system (NSS) and the normal diet implemented by the hospital will be evaluated against the group of patients receiving only the diet, using clinical examination, laboratory and cabinet tests during their hospital stay.

Statistical analysis: for independent groups with normal distribution, Student's T will be applied. If the distribution does not meet normality criteria, a Mann Whitney U will be performed; Two-way ANOVA will be applied to monitor the groups over time with normal distribution. If the distribution does not meet normality criteria, a Friedman test will be performed, in both cases post hoc tests will be performed. The results will be analyzed using version 6 of the Graphpad Prism software.

DETAILED DESCRIPTION:
Patients in the COVID-19 area, who are treated at the ISSEMYM Toluca Arturo Montiel Rojas Medical Center, located in Paseo Tollocan, Av. Baja Velocidad km 575, Barrio de Sta Clara, Toluca de Lerdo, México; both sexes, with the presence of comorbidities (type 2 DM, SAH, overweight or obesity BMI <35) and in stage III of the disease.

Consecutive cases. With systematic randomized allocation using a sequence of random numbers built with the Excel program divided into two groups. Once the participants of the COVID-19 area have been selected, patients and / or family members will be spoken to to explain the protocol and obtain the signatures of the letters of informed consent. Assignment to the research group will be carried out randomly.

Once the patients have been admitted to the study, the following will be carried out: test of COVID-19 by means of PCR, thorax tomography, complete clinical history, Mini Nutritional Assessment (MNA), food diary, list of clinical variables designed by us, complete blood count, coagulation profile, serum electrolytes, blood chemistry (6-elements), lipidic profile, liver function tests, ferritin, fibrinogen, C-reactive protein, procalcitonin and D-dimer. Anthropometric measurements will also be carried out (height, weight, BMI, muscle mass %, fat % and visceral fat%).

The follow-up will be carried out daily for 21 days or earlier, if they are discharged from the hospital due to improvement in the evolution, at that moment the patient concludes the study. The following points will be supervised, recording the information in files and photos, since the hospital security protocol does not allow to extract stationery from the COVID-19 area:

1. Application and consumption of NSS supplementation as appropriate.
2. Morning and evening vital signs.
3. Daily clinical evaluation (It includes variables such as oxygen flow, activity level, integrity of the hair, skin and nails, evaluation of the sense of taste and smell, pain, gastrointestinal symptoms, bowel movements, prescribed medications, mood, among others).
4. Anthropometric measurements using a scale every 2 days (only if the patient is stable and can maintain balance).
5. Food diaries of each patient.
6. Laboratory studies every 3 days (previously mentioned).

In the same way, the following will be taken into account: the number of days hospitalized, number of patients who progress to ventilation, number of patients who die, number of patients who are extubated and number of days after extubation.

A descriptive analysis will be carried out for each continuous variable. These variables will be expressed as mean ± standard deviation and standard error. It will be done according to the distribution of the data; For independent groups with a normal distribution, Student's T will be applied. If the distribution does not meet normality criteria, a Mann Whitney U will be performed; For the follow-up of dependent groups with normal distribution, two-way ANOVA will be applied. If the distribution does not meet normality criteria, a Friedman test will be performed, in both cases post hoc tests will be performed, taking into account that a significant value of p of < 0.05. The results will be analyzed using version 6 of the Graphpad Prism software.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ISSEMYM Toluca Medical Center "Arturo Montiel Rojas ", diagnosed with COVID-19 confirmed by PCR.
* Patients in need of supplemental O2 with nasal prongs or reservoir-mask for satO2 <90% and respiratory distress.
* With concomitant diseases such as cardiovascular disease, diabetes mellitus 2, hypertension, overweight or obesity BMI <35.
* Both sexes.
* Over 30 years old.
* The patient tolerate oral feeding.
* Signing of the letter of informed consent.

Exclusion Criteria:

* Detachment from treatment.
* Admission to the ICU for any reason.
* Patients who do not tolerate the oral route.
* Reactions to treatment that compromise the health of patients.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernado Leal Martínez, Ph.D, Principal Investigator — Anahuac University
Locations (1):
- ISSEMYM "Arturo Montiel Rojas" Medical Center, Toluca, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hummel T, Landis BN, Huttenbrink KB. Smell and taste disorders. GMS Curr Top Otorhinolaryngol Head Neck Surg. 2011;10:Doc04. doi: 10.3205/cto000077. Epub 2012 Apr 26. PMID 22558054
- [Result] Mortazavi H, Shafiei S, Sadr S, Safiaghdam H. Drug-related Dysgeusia: A Systematic Review. Oral Health Prev Dent. 2018;16(6):499-507. doi: 10.3290/j.ohpd.a41655. PMID 30574604
- [Result] Chumpitazi BP, Self MM, Czyzewski DI, Cejka S, Swank PR, Shulman RJ. Bristol Stool Form Scale reliability and agreement decreases when determining Rome III stool form designations. Neurogastroenterol Motil. 2016 Mar;28(3):443-8. doi: 10.1111/nmo.12738. Epub 2015 Dec 21. PMID 26690980
- [Result] Seo AY, Kim N, Oh DH. Abdominal bloating: pathophysiology and treatment. J Neurogastroenterol Motil. 2013 Oct;19(4):433-53. doi: 10.5056/jnm.2013.19.4.433. Epub 2013 Oct 7. PMID 24199004
- [Result] Silva DAS, de Lima TR, Tremblay MS. Association between Resting Heart Rate and Health-Related Physical Fitness in Brazilian Adolescents. Biomed Res Int. 2018 Jun 28;2018:3812197. doi: 10.1155/2018/3812197. eCollection 2018. PMID 30050928
- [Result] Moskowitz A, Patel PV, Grossestreuer AV, Chase M, Shapiro NI, Berg K, Cocchi MN, Holmberg MJ, Donnino MW; Center for Resuscitation Science. Quick Sequential Organ Failure Assessment and Systemic Inflammatory Response Syndrome Criteria as Predictors of Critical Care Intervention Among Patients With Suspected Infection. Crit Care Med. 2017 Nov;45(11):1813-1819. doi: 10.1097/CCM.0000000000002622. PMID 28759474
- [Result] Holvoet E, Vanden Wyngaert K, Van Craenenbroeck AH, Van Biesen W, Eloot S. The screening score of Mini Nutritional Assessment (MNA) is a useful routine screening tool for malnutrition risk in patients on maintenance dialysis. PLoS One. 2020 Mar 4;15(3):e0229722. doi: 10.1371/journal.pone.0229722. eCollection 2020. PMID 32130271
- [Result] Nuttall FQ. Body Mass Index: Obesity, BMI, and Health: A Critical Review. Nutr Today. 2015 May;50(3):117-128. doi: 10.1097/NT.0000000000000092. Epub 2015 Apr 7. PMID 27340299
- [Result] Babiker A, Al Dubayee M. Anti-diabetic medications: How to make a choice? Sudan J Paediatr. 2017;17(2):11-20. doi: 10.24911/SJP.2017.2.12. PMID 29545660
- [Result] Pahan K. Lipid-lowering drugs. Cell Mol Life Sci. 2006 May;63(10):1165-78. doi: 10.1007/s00018-005-5406-7. PMID 16568248
- [Result] Ghoshal K, Bhattacharyya M. Overview of platelet physiology: its hemostatic and nonhemostatic role in disease pathogenesis. ScientificWorldJournal. 2014 Mar 3;2014:781857. doi: 10.1155/2014/781857. eCollection 2014. PMID 24729754
- [Result] Selders GS, Fetz AE, Radic MZ, Bowlin GL. An overview of the role of neutrophils in innate immunity, inflammation and host-biomaterial integration. Regen Biomater. 2017 Feb;4(1):55-68. doi: 10.1093/rb/rbw041. PMID 28149530
- [Result] Hayiroglu MI, Cinar T, Tekkesin AI. Fibrinogen and D-dimer variances and anticoagulation recommendations in Covid-19: current literature review. Rev Assoc Med Bras (1992). 2020 Jun;66(6):842-848. doi: 10.1590/1806-9282.66.6.842. Epub 2020 Jul 20. PMID 32696883
- [Result] Knovich MA, Storey JA, Coffman LG, Torti SV, Torti FM. Ferritin for the clinician. Blood Rev. 2009 May;23(3):95-104. doi: 10.1016/j.blre.2008.08.001. Epub 2008 Oct 2. PMID 18835072
- [Result] Liu F, Li L, Xu M, Wu J, Luo D, Zhu Y, Li B, Song X, Zhou X. Prognostic value of interleukin-6, C-reactive protein, and procalcitonin in patients with COVID-19. J Clin Virol. 2020 Jun;127:104370. doi: 10.1016/j.jcv.2020.104370. Epub 2020 Apr 14. PMID 32344321
- [Result] Kashani K, Rosner MH, Ostermann M. Creatinine: From physiology to clinical application. Eur J Intern Med. 2020 Feb;72:9-14. doi: 10.1016/j.ejim.2019.10.025. Epub 2019 Nov 8. PMID 31708357
- [Result] Wang H, Ran J, Jiang T. Urea. Subcell Biochem. 2014;73:7-29. doi: 10.1007/978-94-017-9343-8_2. PMID 25298336
- [Result] Musso CG, Alvarez-Gregori J, Jauregui J, Macias-Nunez JF. Glomerular filtration rate equations: a comprehensive review. Int Urol Nephrol. 2016 Jul;48(7):1105-10. doi: 10.1007/s11255-016-1276-1. Epub 2016 Apr 6. PMID 27052619
- [Result] Hamade B, Huang DT. Procalcitonin: Where Are We Now? Crit Care Clin. 2020 Jan;36(1):23-40. doi: 10.1016/j.ccc.2019.08.003. Epub 2019 Oct 21. PMID 31733680
- [Result] Driscoll JJ, Rixe O. Overall survival: still the gold standard: why overall survival remains the definitive end point in cancer clinical trials. Cancer J. 2009 Sep-Oct;15(5):401-5. doi: 10.1097/PPO.0b013e3181bdc2e0. PMID 19826360
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Shakoor H, Feehan J, Al Dhaheri AS, Cheikh Ismail L, Ali HI, Alhebshi SH, Apostolopoulos V, Stojanovska L. Role of vitamin D supplementation in aging patients with COVID-19. Maturitas. 2021 Oct;152:63-65. doi: 10.1016/j.maturitas.2021.03.006. Epub 2021 Mar 16. No abstract available. PMID 33757717
- See also: BMI Classification Percentile And Cut Off Points — http://www.ncbi.nlm.nih.gov/books/NBK541070/
- See also: Diabetes Mellitus Type 2 — http://www.ncbi.nlm.nih.gov/books/NBK513253/
- See also: Cardiovascular Disease — http://www.ncbi.nlm.nih.gov/books/NBK535419/
- See also: Hyperlipidemia — http://www.ncbi.nlm.nih.gov/books/NBK559182/
- See also: Dyspnea — http://www.ncbi.nlm.nih.gov/books/NBK499965/
- See also: Chapter 84: Nausea and Vomiting — http://www.ncbi.nlm.nih.gov/books/NBK410/
- See also: Acute Headache — https://www.ncbi.nlm.nih.gov/books/NBK554510/
- See also: Myalgia — http://www.ncbi.nlm.nih.gov/medgen/68541
- See also: Diarrhea — http://www.ncbi.nlm.nih.gov/books/NBK448082/
- See also: Physiology, Respiratory Rate — http://www.ncbi.nlm.nih.gov/books/NBK537306/
- See also: Oxygen Saturation — http://www.ncbi.nlm.nih.gov/books/NBK525974/
- See also: How is body temperature regulated and what is fever? — http://www.ncbi.nlm.nih.gov/books/NBK279457/
- See also: Oxygen Administration — https://www.ncbi.nlm.nih.gov/books/NBK551617/
- See also: Antihypertensive Medications — https://www.ncbi.nlm.nih.gov/books/NBK554579/
- See also: Antibiotics — https://www.ncbi.nlm.nih.gov/books/NBK535443/
- See also: Antacids — https://www.ncbi.nlm.nih.gov/books/NBK526049/
- See also: Nonsteroidal Anti-inflammatory Drugs (NSAIDs) — https://www.ncbi.nlm.nih.gov/books/NBK547742/
- See also: Chapter 151: Hemoglobin and Hematocrit — https://www.ncbi.nlm.nih.gov/books/NBK259/
- See also: Chapter 152: Red Cell Indices — https://www.ncbi.nlm.nih.gov/books/NBK260/
- See also: Histology, White Blood Cell — https://www.ncbi.nlm.nih.gov/books/NBK563148/
- See also: Blood Glucose Monitoring — https://www.ncbi.nlm.nih.gov/books/NBK555976/
- See also: Physiology, Cholesterol — https://www.ncbi.nlm.nih.gov/books/NBK470561/
- See also: Alanine Amino Transferase — https://www.ncbi.nlm.nih.gov/books/NBK559278/
- See also: Chapter 101: Serum Albumin and Globulin — https://www.ncbi.nlm.nih.gov/books/NBK204/
- See also: Calories: Total Macronutrient Intake, Energy Expenditure, and Net Energy Stores — https://www.ncbi.nlm.nih.gov/books/NBK218769/

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Patients who received medical treatment indicated by the hospital and a diet established by the hospital nutrition department of the ISSEMyM Toluca Arturo Montiel Rojas Medical Center.
- Intervention Group: Patients who received medical treatment indicated by the hospital and a diet established by the hospital nutrition department of the ISSEMyM Toluca Arturo Montiel Rojas Medical Center.
  Also it received the Nutritional support system (NSS), which consists of:
  1. 10 mg of cyanocobalamin, 100 mg of thiamin and 100 mg of pyridoxine administered intramuscularly every 24 hours for the first 5 days.
  2. Probiotics Saccharomyces Boulardii (SB) 50 million CFU daily for 6 days orally.
  3. One packet of NSS orally after morning meals and another after evening meals, mixed with 400 ml of water each, during the whole intervention for a maximum of 21 days.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 40 | 40
Completed | 33 | 39
Not Completed | 7 | 1
Not completed — Death | 7 | 1

BASELINE CHARACTERISTICS:
Population: all participants enrolled in the study, a total of 80 patients were compared.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Time elapsed from the birth of a living being to the moment the calculation is made. Based on an official ID. A number between 30 and 75.
  years | 53.9 (10.3) | 51.5 (11.4) | 52.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Set of peculiarities that characterize the individuals of a species, dividing them into male and female, and make possible a reproduction characterized by genetic diversification. Based on an official ID. Categories: 1. Female 2. Male.
  Participants
    Female | 13 | 15 | 28
    Male | 27 | 25 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 40 | 80
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Place where the sample was collected
  participants
    Mexico | 40 | 40 | 80
Overweight [Count of Participants; unit: Participants] — BMI greater than or equal to 25 to 29.9 kg/m^2. The patient is weighed in the baseline period within the physical examination (Approximate duration of 2 minutes). A bioimpedance scale was used.
  Participants | 38 | 36 | 74
Obesity Type I-II [Count of Participants; unit: Participants] — The number of patients who presented BMI 30-39.9 kg/m^2. A bioimpedance scale was used.
  Participants | 14 | 13 | 27
Diabetes Mellitus 2 [Count of Participants; unit: Participants] — the number of patients who were already diagnosed and receiving treatment with hypoglycemic agents and/or insulin prior to the start of the study
  Participants | 13 | 11 | 24
Cardiovascular Disease and/or Hypertension [Count of Participants; unit: Participants] — Cardiovascular disease, also known as heart disease, refers to the following 4 entities: coronary artery disease (CAD) which is also referred to as coronary heart disease (CHD), cerebrovascular disease, peripheral artery disease (PAD), and aortic atherosclerosis. Hypertension is a persistent BP reading of 140/90mmHg or more. It is asked in the baseline period within the clinical history (approximately 10 minutes). Diagnosis is not made upon admission because the physiological stress caused by COVID-19 increases BP and can lead to false positives.
  Participants | 17 | 10 | 27
Hyperlipidemia [Count of Participants; unit: Participants] — Hyperlipidemia is low-density lipoprotein (LDL), total cholesterol, triglyceride levels, or lipoprotein levels greater than the 90th percentile in comparison to the general population, or an HDL level less than the 10th percentile when compared to the general population. It is asked in the baseline period within the medical history (The elaboration of the medical history lasts approximately 10 minutes)
  Participants | 11 | 7 | 18
Number of Participants with Gastrointestinal Disease [Count of Participants; unit: Participants] — Any disease between the esophagus and rectum was considered
  1. Present. 2. Absent. It is asked in the baseline period within the medical history.
  Participants | 14 | 13 | 27
Total Risk Factors [Mean (Standard Deviation); unit: number of risk factors] — Number of diseases present considering: Overweight or obesity, DM2, cardiovascular disease, hyperlipidemia and gastrointestinal disease. Diseases that are in the non-inclusion criteria are not considered. The summation is made in the baseline period within the clinical history (The elaboration of the clinical history takes approximately 10 minutes).
  number of risk factors | 2.92 (1.42) | 2.57 (1.35) | 2.75 (1.39)
Number of Participants with Dyspnea [Count of Participants; unit: Participants] — Commonly referred to as shortness of breath, is the subjective sensation of uncomfortable breathing comprised of various sensations of varying intensity.
  1. Present, 2. Absent. It is asked in the baseline period within the medical history (The elaboration of the medical history lasts approximately 10 minutes)
  Participants | 24 | 26 | 50
Nausea and Vomiting [Count of Participants; unit: Participants] — Vomiting, or emesis, is the forceful retrograde expulsion of gastric contents from the body. Nausea is the unpleasant sensation that precedes vomiting. It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 6 | 7 | 13
Hyposmia [Count of Participants; unit: Participants] — Hyposmia refers to a reduced ability to smell. It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 12 | 15 | 27
Dysgeusia [Count of Participants; unit: Participants] — Dysgeusia is an unpleasant alteration in taste. It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 18 | 20 | 38
Number of Participants with Headache [Count of Participants; unit: Participants] — Pain located in any part of the head.
  1. Present, 2. Absent It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 26 | 29 | 55
Number of Participants with Myalgia [Count of Participants; unit: Participants] — Pain in muscle.
  1. Present, 2. Absent It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 32 | 30 | 62
Number of Participants with Diarrhea [Count of Participants; unit: Participants] — Diarrhea is described as three or more loose or watery stools a day. 1. Present, 2. Absent It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 18 | 12 | 30
Number of Participants with Anorexia [Count of Participants; unit: Participants] — Occurs when the desire to eat is reduced. 1. Present, 2. Absent It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 20 | 21 | 41
Total of symptoms [Mean (Standard Deviation); unit: number of symptoms] — Summation of symptoms including dyspnea, nausea or vomiting, hyposmia, dysgeusia, headache, myalgia, diarrhea, and lack of appetite. The summation is made in the baseline period within the clinical history (The elaboration of the clinical history takes approximately 10 minutes).
  number of symptoms | 7.05 (2.11) | 6.8 (2.23) | 6.92 (2.16)
Bristol scale "normal" (T3-4) [Count of Participants; unit: Participants] — The Bristol Stool Form Scale categorizes stools into one of seven stool types ranging from type 1 (hard lumps) to type 7 (watery diarrhea).
  Type 3 and 4 were considered "Normal". The patient is asked the consistency of the stool in the baseline period (duration approximately 10 minutes).
  Participants | 9 | 5 | 14
Number of defecations [Mean (Standard Deviation); unit: Number of defecations per day] — The patient is asked the number of times he defecates daily, in the baseline period (duration approximately 10 minutes).
  Number of defecations per day | 0.54 (0.6) | 0.52 (0.73) | 0.53 (0.66)
Number of Participants with Abdominal Distension [Count of Participants; unit: Participants] — Is a visible increase in abdominal girth.
  1. Present, 2. Absent. The patient is explored in the baseline period (duration approximately 10 minutes).
  Participants | 28 | 28 | 56
Breathing Frequency [Mean (Standard Deviation); unit: breaths per minute] — The number of breaths per minute (bpm). The patient is explored in the baseline period (duration approximately 10 minutes).
  breaths per minute | 21.18 (3.01) | 21.48 (3.01) | 21.32 (2.99)
Oxygen Saturation [Mean (Standard Deviation); unit: oxygen saturation percentage] — Measures how much hemoglobin is currently bound to oxygen compared to how much hemoglobin remains unbound. A pulse oximeter can measure oxygen saturation. It is a noninvasive device placed over a person's finger. It measures light wavelengths to determine the ratio of the current levels of oxygenated hemoglobin to deoxygenated hemoglobin. It is evaluated in the baseline period within the clinical history (approximately 10 minutes).
  oxygen saturation percentage | 92.73 (4.17) | 94 (3.18) | 93.36 (3.74)
Resting Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Heart rate (HR) reflects the number of contractions of the ventricles per unit time and fluctuates substantially with variations in systemic demand for oxygen. Resting heart rate (RHR) monitoring is a simple and noninvasive clinical method. It is evaluated in the baseline period within the clinical history (approximately 10 minutes).
  beats per minute | 70.7 (15.4) | 75.5 (9.88) | 73.07 (13.07)
Body Temperature (ºC) [Mean (Standard Deviation); unit: degrees Celsius (ºC)] — Because we cannot measure the temperature inside these organs, temperature is taken on parts of the body that are more accessible.Balance between the production of heat by the body and its loss. Measurement using an infrared thermometer. Units of measure degrees centigrade. Average taken morning and evening measurements. It is evaluated in the baseline period within the clinical history (approximately 10 minutes).
  degrees Celsius (ºC) | 36.27 (0.73) | 36.25 (0.62) | 36.25 (0.67)
Liters of Supplemental Oxygen [Mean (Standard Deviation); unit: L/min] — Supplemental oxygen that is above the amount found in the atmosphere without alteration, delivered to the patient by nasal cannula or O2 mask. It is evaluated in the baseline period within the clinical history (approximately 10 minutes).
  L/min | 5.9 (3.82) | 6 (3.29) | 5.97 (3.54)
qSOFA Score [Mean (Standard Deviation); unit: units on a scale] — Quick-Sequential Organ Failure Assessment (qSOFA) score gives 0 to 3 points. ≥2 in the setting of suspected infection had a high predicted in-hospital mortality rate and could be considered septic. It is evaluated in the baseline period within the clinical history (approximately 10 minutes).
  units on a scale | 0.425 (0.59) | 0.65 (0.62) | 0.53 (0.61)
MNA (Mini Nutritional Assessment) Score [Mean (Standard Deviation); unit: units on a scale] — The Mini Nutritional Assessment score is a validated nutritional screening that identifies malnutrition or risk of malnutrition.
  The tool consists of a short screening form of 18 items in the long version and 6 items in the short version; with score ranges between 0 minimum and 30 maximum, questions A-E should be answered and the sum of the total score should be ranked.
  * 12 to 30 points: indicates adequate nutrition and does not require nutritional intervention.
  * 8 and 11 ponis indicates risk of malnutrition.
  * 7 or less points indicates malnutrition. maximum score 14 points.
  units on a scale | 11.13 (2.26) | 11.38 (1.65) | 11.25 (1.97)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — The body mass index (BMI) is the metric currently in use for defining anthropometric height/weight characteristics in adults and for classifying (categorizing) them into groups.
  Normal weight - BMI greater than or equal to 18.5 to 24.9 kg / m ^ 2. It is evaluated in the baseline period within the clinical history (approximately 10 minutes).
  kg/m^2 | 29.35 (3.89) | 29.98 (4.07) | 29.66 (3.97)
Hydric Balance [Mean (Standard Deviation); unit: milliliters] — Hydric balance quantified in milliliters. It is evaluated in the baseline period within the clinical history (approximately 10 minutes).
  milliliters | -203.4 (966) | -301.5 (1167) | -254.1 (1056)
Antihypertensive medication [Count of Participants; unit: Participants] — There are multiple classes of antihypertensive medications used for the treatment of HTN like: Thiazide-type diuretics, Calcium channel blockers, Angiotensin-converting enzyme (ACE) inhibitors and angiotensin II receptor blockers (ARBs), Beta-blockers, etc. It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 13 | 9 | 22
Antidiabetics medication [Count of Participants; unit: Participants] — The main goals of Anti-diabetes therapy are to reduce symptoms of hyperglycaemia and to reduce the risk of long-term complications of diabetes. We include insulins, GLP-1 agonists, Biguanides, Sulphonylureas, Thiazolidinediones, 'Gliptins', α-glucosidase inhibitors, SGLT2 inhibitor, etc. It is asked in the baseline period within the medical history (approximately 10 minutes).
  Participants | 9 | 11 | 20
Antilipids medication [Count of Participants; unit: Participants] — Most of the lipid-lowering drugs are classified mainly into two groups: statins and fibrates. It is asked in the baseline period within the medical history (The elaboration of the medical history lasts approximately 10 minutes).
  Participants | 3 | 3 | 6
Antibiotics medication [Count of Participants; unit: Participants] — Antibiotics are compounds that target bacteria and, thus, are intended to treat and prevent bacterial infections.
  It is asked in the baseline period within the medical history (The elaboration of the medical history lasts approximately 10 minutes).
  Participants | 1 | 4 | 5
Antiacids [Count of Participants; unit: Participants] — Antacids are a combination of various compounds with various salts of calcium, magnesium, and aluminum as the active ingredients. The antacids act by neutralizing the acid in the stomach and by inhibiting pepsin, which is a proteolytic enzyme.
  it is asked in the baseline period within the medical history (The elaboration of the medical history lasts approximately 10 minutes).
  Participants | 6 | 6 | 12
NSAIDs medication [Count of Participants; unit: Participants] — NSAIDs are a class of medications used to treat pain, fever, and other inflammatory processes.
  It is asked in the baseline period within the medical history if the patient is taking any antiacid (The elaboration of the medical history lasts approximately 10 minutes).
  Participants | 8 | 12 | 20
Hemoglobin [Mean (Standard Deviation); unit: g/dL] — Hemoglobin (Hb) is the protein contained in red blood cells that is responsible for delivery of oxygen to the tissues. The amount of hemoglobin in whole blood is expressed in grams per deciliter (g/dl). The normal Hb level for males is 14 to 18 g/dl; that for females is 12 to 16 g/dl.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  g/dL | 15.53 (2.22) | 15.54 (2.08) | 15.53 (2.14)
Mean Corpuscular Hemoglobin Concentration [Mean (Standard Deviation); unit: g/dL] — MCHC indicates the amount of hemoglobin per unit volume. In contrast to MCH, MCHC correlates the hemoglobin content with the volume of the cell. It is expressed as g/dl of red blood cells or as a percentage value. The normal values for MCHC are 34 ± 2 g/dl.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  g/dL | 33.39 (1.4) | 33.46 (1.17) | 33.42 (1.28)
Platelets [Mean (Standard Deviation); unit: 10^3 platelets / μL] — Platelets are small anucleate cell fragments that circulate in blood playing crucial role in managing vascular integrity and regulating hemostasis. Platelets are also involved in the fundamental biological process of chronic inflammation associated with disease pathology. The normal platelet count is (150-400) × 10^3 per microliter of blood.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  10^3 platelets / μL | 222.2 (53.93) | 248.4 (139.9) | 235.3 (106.1)
Leukocytes [Mean (Standard Deviation); unit: 10^3 leukocytes / μL] — White blood cells, or leukocytes, are part of the immune system participating in both the innate and humoral immune responses. They circulate in the blood and mount inflammatory and cellular responses to injury or pathogens. The normal range of values for white blood cells is 4,000 to 11,000/mL.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  10^3 leukocytes / μL | 8.97 (4.15) | 8.46 (4.36) | 8.72 (4.23)
Neutrophils [Mean (Standard Deviation); unit: percentage] — Neutrophils are polymorphonuclear lymphocytes that reside mainly in the peripheral vasculature. The standard circulating neutrophil count is above 1.5 x 10/L.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  percentage | 83.5 (8.87) | 80.78 (9.29) | 82.14 (9.12)
Glycemia [Mean (Standard Deviation); unit: mg/dL] — Normal range: 4 to 6 mmol or about 72 to 108 mg/dL. Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  mg/dL | 135.4 (59.39) | 134.8 (58.83) | 135.12 (58.73)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] — Cholesterol contributes to the structural makeup of the membrane as well as modulates its fluidity. Cholesterol functions as a precursor molecule in the synthesis of vitamin D, steroid hormones (e.g., cortisol and aldosterone and adrenal androgens), and sex hormones (e.g., testosterone, estrogens, and progesterone). Cholesterol is also a constituent of bile salt used in digestion to facilitate absorption of fat-soluble vitamins A, D, E, and K.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  mg/dL | 142.8 (42.82) | 135 (23.53) | 138.98 (34.65)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Triglycerides are fatty acid esters of glycerol and represent the main lipid component of dietary fat and fat depots of animals. The general population's ideal triglyceride level is less than 150 mg/dL.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  mg/dL | 147.5 (58.92) | 132.8 (37.39) | 140.2 (49.6)
AST [Mean (Standard Deviation); unit: U/L] — Serum hepatic enzyme. Normal serum aspartate aminotransferase (AST) is 0 to 35 U/L.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  U/L | 48.06 (28.81) | 46.4 (49.65) | 47.2 (40.3)
ALT [Mean (Standard Deviation); unit: U/L] — Serum hepatic enzyme. Normal serum alanine aminotransferase (ALT) is 7-56 U/L. Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  U/L | 47.69 (31.9) | 50.44 (50.88) | 49.06 (42.21)
Albumin [Mean (Standard Deviation); unit: g/dL] — Albumin is the most abundant circulating protein found in plasma. The normal serum albumin is 3.5 to 5.0 g/dl.
  Laboratory samples are taken in the baseline period. The time to obtain the blood sample is approximately 1 minute.
  g/dL | 3.53 (0.44) | 3.57 (0.41) | 3.55 (0.42)
Ferritin [Mean (Standard Deviation); unit: ng/ml] — An iron storage protein. Is the primary iron storage mechanism and is critical to iron homeostasis. Reference ranges for serum ferritin vary across laboratories, but levels of 30 to 300 ng/ml are considered normal for men, and 10-200 ng/ml for women.
  Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  ng/ml | 1070 (899.3) | 1270 (1142) | 1167 (1022)
Fibrinogen [Mean (Standard Deviation); unit: mg/dl] — Is one of the acute phase proteins, is synthesized in high quantity by the liver in response to IL-1 and IL-6 derived stimulation, as well as is involved in fibrin formation as the last step of a triggered coagulation activity.
  Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  mg/dl | 592.2 (170.4) | 607.4 (162.9) | 600 (165.3)
CRP [Mean (Standard Deviation); unit: mg/l] — Is a non-specific acute-phase protein induced by IL-6 in the liver and a sensitive biomarker of inflammation, infection, and tissue damage.
  Laboratory samples are taken in the baseline period the time to obtain the blood sample is approximately 1 minute.
  mg/l | 157.3 (106.7) | 135.3 (94.92) | 146.3 (100.9)
D dimer [Mean (Standard Deviation); unit: μg/ml] — Is the soluble plasmin-mediated degradation product of fibrin, which is produced after activation of coagulation and fibrinolysis.
  Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  μg/ml | 291.2 (179.9) | 444.9 (954.9) | 368 (686.4)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dl] — Is the end product of creatine and creatine phosphate metabolism. Is a nitrogenous organic acid that is generated predominantly in the kidney and liver, and to some extent in the pancreas, using three amino acids, glycine, arginine, and methionine. Serum creatinine level for men with normal kidney function is approximately 0.6 to 1.2mg/dL and between 0.5 to 1.1 mg/dL for women.
  Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  mg/dl | 0.88 (0.31) | 0.86 (0.22) | 0.87 (0.27)
Urea [Mean (Standard Deviation); unit: mg/dl] — Is generated by the urea cycle enzymes, which are mainly in the liver but are also ubiquitously expressed at low levels in other tissues. As a terminal product, is subsequently excreted out of the organism after generation. The normal range of urea nitrogen in blood or serum is 5 to 20 mg/dl.
  Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  mg/dl | 33.95 (15.84) | 32.95 (10.78) | 33.42 (13.47)
Blood urea nitrogen (BUN) [Mean (Standard Deviation); unit: mg/dl] — Clinicians usually use blood urea nitrogen (BUN) to measure the amount of nitrogen coming from urea in the blood as an index of renal function. The normal range of urea nitrogen in blood or serum is 5 to 20 mg/dl.
  Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  mg/dl | 15.87 (7.39) | 15.43 (5.02) | 15.65 (6.29)
Glomerular filtration rate (GFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Glomerular filtration rate (GFR) is classically used just for evaluating individual's kidney function and for scoring disease stages in chronic kidney disease (CKD) patients. Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  mL/min/1.73 m^2 | 90.15 (20.2) | 93.59 (17.4) | 91.84 (18.82)
Procalcitonin [Mean (Standard Deviation); unit: μg/L] — Is a protein that consists of 116 amino acids and is the peptide precursor of calcitonin. Is a biomarker generally elevated in bacterial infections but not viral and it is a guidance for physicians to evaluate the decreasing antibiotic use in critically ill patients. Serum PCT concentration in healthy individuals is typically <0.1 μg/L.
  Laboratory samples are taken in the baseline period and the time to obtain the blood sample is approximately 1 minute.
  μg/L | 0.364 (0.6) | 0.18 (0.188) | 0.27 (0.45)
basal energy intake [Mean (Standard Deviation); unit: kilocalories] — One kilocalorie (equivalent to 4.184 kJ) is the amount of heat required to raise the temperature of 1 kg of water 1°C (e.g., from 15 to 16°C) at standard atmospheric pressure (760 mm Hg). Food diaries are made that are subsequently analyzed by a nutritionist. The realization of the food diary is done 3 times a day after the meal (5 minutes each approximately)
  kilocalories | 1411 (46.2) | 1376 (36.3) | 1393.5 (43.3)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival, the total number of patients included in the study and completed a 40-day follow-up.
Time Frame: 40 days.
Population: the total number of patients who were enrolled and included in the study and who survived or not at the end of follow-up at day 40.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 33 | 39
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; The total number of patients who did or did not survive to day 40 of follow-up; Test type: Other — Kaplan-Meier method for overall survival; p = 0.027, Log Rank

2. Primary Outcome: Overall Mortality at Day 40
Description: Total number of patients who died before day 40 of follow-up.
Time Frame: 40 days.
Population: total number of patients who were enrolled in the study and died prior to day 40 of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 7 | 1

3. Secondary Outcome: Survival in Intubated Patients at Day 40
Description: Total number of patients who were intubated, extubated, discharged and completes the 40 day follow-up
Time Frame: 40 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 7 | 3
Participants | 2 | 2
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; the total number of patients who were intubated and survived at the end of day 40 follow-up; Test type: Other — Kaplan-Meier method; p = 0.495, Log Rank

4. Secondary Outcome: Mortality in Intubated Patients at Day 40
Description: Patients who were intubated during their hospital stay and died before completing follow-up on day 40.
Time Frame: 40 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 7 | 3
Participants | 5 | 1

5. Secondary Outcome: Progression to Mechanical Ventilation Assistance
Description: total number of patients included in the study who progressed to mechanical ventilation during the first 10 days of hospital stay.
Time Frame: 10 days.
Population: Proportion of patients from control group and intervention group were analyzed with the Kaplan-Meier method comparing both groups to MVA progression
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 7 | 3
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; total number of patients included in the study who progressed to mechanical ventilation during the first 10 days of hospital stay; Test type: Other — Kaplan-Meier method; p = 0.186, Log Rank

6. Secondary Outcome: Participants With Normal Bristol Scale at Day 3
Description: The Bristol Stool Form Scale categorizes stools into one of seven stool types ranging from type 1 (hard lumps) to type 7 (watery diarrhea). Type 3 and 4 were considered "Normal".
Time Frame: day 3
Population: Intergroup analysis between the control group and the intervention group, measured at day 3 of hospital stay . Deceased patients were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 24 | 31
Participants | 8 | 13
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Intergroup analysis between the control group and the intervention group, measured at day 3 of hospital stay. It was categorized as follows: 1. normal bristol scale at day 3; 2. abnormal bristol scale at day 3; Test type: Superiority — Fisher exact test; p = 0.35, Fisher Exact

7. Secondary Outcome: Hidric Balance on Day 3
Description: The ratio between the water assimilated into the body and that lost from the body, in milliliters.
Time Frame: It is evaluated on day 3 of hospital stay (duration approximately 10 minutes).
Population: Intergroup analysis between the control group and the intervention group for different parameters, measured at day 3 of hospital stay . Deceased patients were excluded.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 18
milliliters | 123.4 (453.8) | 456.6 (485.5)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Intergroup analysis between the control group and the intervention group, measured at day 3 of hospital stay . Deceased patients were excluded; Test type: Superiority; p = 0.043, t-test, 1 sided

8. Secondary Outcome: Oxigen Saturation >90% on Day 3
Description: the total number of patients with oxygen saturation >90% on day 3 of their hospital stay.
Time Frame: day 3.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Participants | 34 | 37
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Intergroup analysis between the control group and the intervention group for different parameters, measured at day 3 of hospital stay . Deceased patients were excluded; Test type: Superiority; p = 0.241, Fisher Exact

9. Secondary Outcome: PHQ-9 Test
Description: Is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders, includes 9 items, which evaluate the presence of depressive symptoms based on the criteria of the Diagnostic and Statistical Manual of Mental Disorders version 4, during the last 2 weeks, how often the patient presented depressive symptoms. According to the sum of the score obtained, the following 4 categories will be considered: 0-4 minimum existence or absence of depressive symptoms; 5-9 = mild depressive symptoms; 10-14 = moderate depressive symptoms; 15-19 = moderate to severe depressive symptoms; 20-27 = severe depressive symptoms.
Time Frame: baseline and hospital discharge
Population: Intragroup analysis between the control group and the intervention group for different parameters, measured at baseline and at hospital discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 6 | 10
score on a scale
  Baseline | 3.66 (2.5) | 5.3 (3.4)
  Hospital discharge | 1.50 (2.8) | 1.9 (1.4)
Statistical Analysis 1: Comparison: Control Group; Intragroup analysis at the control group, the measurement was performed at baseline and at hospital discharge; Test type: Superiority; p = 0.187, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group; Intragroup analysis at the intervention group, the measurement was performed at baseline and at hospital discharge; Test type: Superiority; p = 0.003, t-test, 2 sided

10. Secondary Outcome: Oxigen Flow (Intragroup)
Description: Difference in oxygen delivery between the baseline period and day 3 of hospital stay in each group.
Time Frame: baseline and day 3
Population: Intragroup and Intergroup analysis between the control group and the intervention group for the difference in oxygen delivery between the baseline period and day 3 of hospital stay in each group.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
Liters (L)
  Baseline | 5.9 (3.8) | 6 (3.2)
  Day 3 | 6 (4.4) | 4.5 (3.5)
Statistical Analysis 1: Comparison: Control Group; Intragroup analysis of the control group in oxygen delivery, the difference between the baseline period and day 3 of hospital stay; Test type: Superiority; p = 0.919, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.014, t-test, 2 sided

11. Secondary Outcome: qSOFA at Day 3
Description: Quick-Sequential Organ Failure Assessment (qSOFA) score gives 0 to 3 points. ≥2 in the setting of suspected infection had a high predicted in-hospital mortality rate and could be considered septic.
Time Frame: Baseline and Day 3
Population: Intragroup analysis of both groups, the difference in the qSOFA measurement at baseline and at day 3 will be analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 0.42 (0.59) | 0.65 (0.62)
  Day 3 | 0.51 (0.57) | 0.43 (0.49)
Statistical Analysis 1: Comparison: Control Group; Intragroup analysis of the control group, the difference in the qSOFA measurement at baseline and at day 3 will be analyzed; Test type: Superiority; p = 0.608, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Intragroup analysis of the intervention group, the difference in the qSOFA measurement at baseline and at day 3 will be analyzed; Test type: Superiority; p = 0.04, t-test, 2 sided

12. Secondary Outcome: Number of Defectations on Day 3
Description: Refers to the subjective sensation of increased abdominal pressure without an increase in abdominal size, the number of defecations were quantified at day 3 and compared between both groups.
Time Frame: Day 3
Population: Intergroup analysis between both groups to evaluate the number of defecations measured at day 3.
Measure: Mean (Standard Deviation); unit: defecations
Groups:
- Intervention Group: Patients who received the nutritional support system (NSS) and the standard diet
  Nutritional support system (NSS): 1.Combination of three B vitamins (B1, B6 and B12) "Neurobion" 10 mg solution for IM injection, One every 24 hours for the first 5 days.
  2.Probiotics Saccharomyces boulardii CNCM I-745 "Floratil". One morning and one evening 250 mg capsule during the first 6 days
  3. One envelope of NSS-1 in the morning and one envelope in the afternoon mixed with 400 ml of water each, contain nutritional support system.
  Conventional nutritional support designed by hospital nutritionists: Diet designed by the nutrition department according to comorbidities and intubation probability. Food will be established according to the provisions of the ISSEMYM Toluca Arturo Montiel Rojas Medical Center.
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 37 | 36
defecations | 0.81 (0.90) | 1.41 (1.13)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Intergroup analysis between both groups to evaluate the number of defecations measured at day 3; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Number of Participants With Distension on Day 3
Description: Is a visible increase in abdominal girth.1. Present, 2. Absent.
Time Frame: Day 3
Population: Intergroup analysis between the control group and the intervention group for different parameters, measured at day 3 of hospital stay. Deceased patients were excluded.
Measure: Number; unit: percent of participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 31 | 31
percent of participants | 51.6 | 19.4
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Intergroup analysis between the control group and the intervention group for different parameters, measured at day 3 of hospital stay. Deceased patients were excluded; Test type: Superiority; p = 0.008, Fisher Exact; the shapiro wilk test was used to analyze the distribution of the data

14. Other Pre Specified Outcome: Saturation Without Supplementary Oxygen
Description: The oxygen saturation without supplementary oxygen is taken at the control appointment 40 days after hospital discharge.
Time Frame: day 40
Population: Intergroup analysis between the control group and the intervention group for different parameters, measured at a complete follow-up of 40 days. Deceased patients were excluded.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 28 | 38
percentage | 90.39 (3.4) | 92.08 (2.5)

15. Other Pre Specified Outcome: Need for Home Oxygen Flow
Description: The need to continue with supplemental oxygen at hospital discharge. Categories: 1. Yes, 2. No.
Time Frame: Day 40
Population: Intragroup analysis between the control group and the intervention group for different parameters, measured at a complete follow-up of 40 days of hospital stay. Deceased patients were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 27 | 39
Participants | 23 | 26
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority — Intergroup analysis between the control group and the intervention group for different parameters, measured at a complete follow-up of 40 days. Deceased patients were excluded; p = 0.078, Fisher Exact

16. Other Pre Specified Outcome: Time of Home Oxigen Use
Description: It is recorded for how many days the treating doctor asked the patients to continue to administer supplemental oxygen after hospital discharge
Time Frame: day 40
Population: Intragroup analysis between the control group and the intervention group for different parameters, measured at a complete follow-up of 40 days. Deceased patients were excluded
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 17 | 23
days | 57.6 (24.6) | 43.8 (16.2)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Intergroup analysis between the control group and the intervention group for different parameters, measured at a complete follow-up of 40 days. Deceased patients were excluded; Test type: Superiority; p = 0.098, t-test, 1 sided

17. Other Pre Specified Outcome: Post Covid Syndrome
Description: Persistence of clinical signs and symptoms that arise after developing COVID-19, and are not explained by an alternative diagnosis. 1. Present. 2. Absent.
Time Frame: Day 40.
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 24 | 34
Participants | 9 | 8
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Intergroup analysis between the control group and the intervention group to analyze the presentation of post covid syndrome at the end of follow-up at day 40; Test type: Other; p = 0.195, Fisher Exact

18. Other Pre Specified Outcome: Weight Decrease
Description: Is defined as at least a 5% reduction in weight from the baseline level.Total number of patients with weight loss at the end of follow-up at day 40
Time Frame: Day 40
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 11 | 18
Participants | 8 | 8
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.135, Fisher Exact

19. Other Pre Specified Outcome: Gastrointestinal Symptoms
Description: Total number of patients with gastrointestinal symptoms at the end of follow-up at day 40.Those symptoms perceived abdominal region (pain, burn, pressure, nausea, vomiting)
Time Frame: Day 40
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 24 | 37
Participants | 4 | 3
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.266, Fisher Exact

20. Other Pre Specified Outcome: Number of Deceased Patients Stratified by Fibrinogen Level.
Description: Association between the presentation of certain laboratory parameters taken at baseline with the overall mortality of discharged patients compared to deceased patients.
Time Frame: Baseline
Population: Association between the presentation of certain laboratory parameters taken at baseline compared to overall mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Fibrinogen <700 mg/dL: Patients with fibrinogen levels <700 mg/dl at baseline and died.
- Fibrinogen >700 mg/dL: Patients with fibrinogen levels > 700 mg/dl at baseline and died.
Arm/Group | Fibrinogen <700 mg/dL | Fibrinogen >700 mg/dL
Number analyzed (Participants) | 61 | 19
Participants | 2 | 6
Statistical Analysis 1: Comparison: Fibrinogen <700 mg/dL vs Fibrinogen >700 mg/dL; Test type: Superiority — Association between the presentation of certain laboratory parameters taken in the baseline period, with te overall mortality of discharge patients in comparison with deceased patients; p = 0.002, Fisher Exact

21. Other Pre Specified Outcome: Number of Deceased Patients Stratified by Procalcitonin Level.
Description: Association between the presentation of certain laboratory parameters taken in the baseline period, with te overall mortality of discharge patients in comparison with deceased patients
Time Frame: Baseline
Population: Association between the presentation of certain laboratory parameters taken at baseline compared to overall mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Procalcitonin <0.5 ng/mL: Patients with procalcitonin levels <0.5 ng/mL at baseline and died.
- Procalcitonin >0.5 ng/mL: Patients with procalcitonin levels >0.5 ng/mL at baseline and died.
Arm/Group | Procalcitonin <0.5 ng/mL | Procalcitonin >0.5 ng/mL
Number analyzed (Participants) | 72 | 8
Participants | 4 | 4
Statistical Analysis 1: Comparison: Procalcitonin <0.5 ng/mL vs Procalcitonin >0.5 ng/mL; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.003, Fisher Exact

22. Other Pre Specified Outcome: Number of Deceased Patients Stratified by Ureic Nitrogen Level
Description: as for outcome 21
Time Frame: Baseline
Population: Association between the presentation of certain laboratory parameters taken at baseline compared to overall mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Ureic Nitrogen <22 mg/dL: Patients with Ureic Nitrogen <22 mg/dL at baseline and died.
- Ureic Nitrogen >22 mg/dL: Patients with Ureic Nitrogen >22 mg/dL at baseline and died.
Arm/Group | Ureic Nitrogen <22 mg/dL | Ureic Nitrogen >22 mg/dL
Number analyzed (Participants) | 71 | 9
Participants | 4 | 4
Statistical Analysis 1: Comparison: Ureic Nitrogen <22 mg/dL vs Ureic Nitrogen >22 mg/dL; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.004, Fisher Exact

23. Other Pre Specified Outcome: Number of Deceased Participants Stratified by RCP Level
Description: as for outcome 21
Time Frame: Baseline
Population: Association between the presentation of certain laboratory parameters taken at baseline compared to overall mortality.
Measure: Count of Participants; unit: Participants
Groups:
- RCP <150 mg/L: Patients with RCP <150 mg/L at baseline and died.
- RCP >150 mg/L: Patients with RCP >150 mg/L at baseline and died.
Arm/Group | RCP <150 mg/L | RCP >150 mg/L
Number analyzed (Participants) | 45 | 35
Participants | 1 | 7
Statistical Analysis 1: Comparison: RCP <150 mg/L vs RCP >150 mg/L; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.011, Fisher Exact

24. Other Pre Specified Outcome: Number of Deceased Participants Stratified by Neutrophils Level
Description: as for outcome 21
Time Frame: Baseline
Population: Association between the presentation of certain laboratory parameters taken at baseline compared to overall mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Neutrophils <80%: Patients with neutrophils <80% at baseline and died
- Neutrophils >80%: Patients with neutrophils >80% at baseline and died
Arm/Group | Neutrophils <80% | Neutrophils >80%
Number analyzed (Participants) | 27 | 53
Participants | 0 | 8
Statistical Analysis 1: Comparison: Neutrophils <80% vs Neutrophils >80%; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.031, Fisher Exact

25. Other Pre Specified Outcome: Number of Deceased Participants Stratified by Leukocytes Level
Description: as for outcome 21
Time Frame: Baseline
Population: Association between the presentation of certain laboratory parameters taken at baseline compared to overall mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Leukocytes <10x10^3/μL: Patients with Leukocytes <10x10^3/μL at baseline and died
- Leukocytes >10x10^3/μL: Patients with Leukocytes >10x10^3/μL at baseline and died
Arm/Group | Leukocytes <10x10^3/μL | Leukocytes >10x10^3/μL
Number analyzed (Participants) | 57 | 23
Participants | 3 | 5
Statistical Analysis 1: Comparison: Leukocytes <10x10^3/μL vs Leukocytes >10x10^3/μL; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.040, Fisher Exact

26. Other Pre Specified Outcome: Number of Deceased Participants Stratified by Urea Level
Description: as for outcome 21
Time Frame: Baseline
Population: Association between the presentation of certain laboratory parameters taken at baseline compared to overall mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Urea <40 mg/dL: Patients with Urea <40 mg/dL at baseline and died
- Urea >40 mg/dL: Patients with Urea >40 mg/dL at baseline and died
Arm/Group | Urea <40 mg/dL | Urea >40 mg/dL
Number analyzed (Participants) | 64 | 16
Participants | 4 | 4
Statistical Analysis 1: Comparison: Urea <40 mg/dL vs Urea >40 mg/dL; Test type: Superiority — [test comment as in outcome 20, analysis 1]; p = 0.047, Fisher Exact

ADVERSE EVENTS:
Time Frame: 40 days.
Description: Adverse Events and All Cause Mortality monitored for 40 days.
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 7/40 | 1/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 5/40
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=40) | Intervention Group (N=40)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
Restriction of resources for laboratory tests, small number of subjects analyzed and restriction of access of measuring instruments to the COVID-19 area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04507867/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04507867/SAP_001.pdf
  • Informed Consent Form (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT04507867/ICF_002.pdf